CLINICAL TRIAL: NCT04445493
Title: EPISODE-PS-COVID: hEad Pulse for Ischemic StrOke DEtection Prehospital Study During the COVID-19 Pandemic
Brief Title: EPISODE-PS-COVID: hEad Pulse for Ischemic StrOke DEtection Prehospital Study During the COVID-19 Pandemic ( EPISODEPSCOVID )
Acronym: EPISODE-PH-COV
Status: Completed | Type: Observational
Sponsor: MindRhythm, Inc. (Industry)
Collaborators: Wayne State University (Other); Western Michigan University (Other)
Responsible Party: Sponsor
Other Study IDs: EPISODE-PH-COVID
Record Dates: First submitted 2020-06-18; First posted 2020-06-24 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-11

CONDITIONS: Stroke, Acute; COVID-19
MeSH Terms: conditions — Stroke; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Device: MindRhythm Harmony: Passive recording of the head pulse
  Interventions: Device: MindRhythm Harmony

INTERVENTIONS:
Device: MindRhythm Harmony — Passive recording of the head pulse
  Other Names: Cranial Accelerometry

SUMMARY:
Prehospital providers encounter patients with suspected stroke frequently. Stroke and COVID-19 are related potentially putting these healthcare workers at risk of COVID-19 infection. In addition, prehospital providers need tools to help triage large vessel stroke patients to comprehensive stroke centers.

DETAILED DESCRIPTION:
This observational prospective study will document COVID-19 status on patients seen in the prehospital environment for suspected stroke. This will provide an estimate of how frequently stroke occurs in stroke and also the exposure risk to providers in this setting.

Additionally, patients will have a headset placed to record their headpulse during the encounter. These measurements will be used to further develop an analytic model used to predict the presence of large vessel occlusion (LVO) stroke. This may help create a device that can be used in the prehospital environment to aid in the trade decision of destination hospital.

ELIGIBILITY:
Inclusion Criteria:

* suspected stroke in the prehospital setting
* patient at risk for COVID-19

Exclusion Criteria:

* scalp laceration
* Patient refusal
* Prisoner, other vulnerable population
* Prehospital provider feels that the recording may interfere with care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are being evaluated in the prehospital environment by Detroit Paramedics/EMTs in whom stroke is suspected and who may be at risk fo COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of COVID-19 infection in suspected stroke population | Through Study Completion, an average of 6 months
Quality head pulse recordings | Through Study Completion, an average 6 months
  Proportion of head pulse studies deemed of high quality for further analysis

CONTACTS AND LOCATIONS:
Overall Officials: James Paxton, MD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Smith WS, Keenan KJ, Lovoi PA. A Unique Signature of Cardiac-Induced Cranial Forces During Acute Large Vessel Stroke and Development of a Predictive Model. Neurocrit Care. 2020 Aug;33(1):58-63. doi: 10.1007/s12028-019-00845-x. PMID 31591693